CLINICAL TRIAL: NCT06329739
Title: Genetics in Parkinson's Disease: Behavioral and Cognitive Outcomes in Patients Undergoing Dopaminergic Treatment
Brief Title: Genetics in Parkinson's Disease: Behavioral and Cognitive Outcomes
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroPsico_Dopa&PD
Record Dates: First submitted 2024-03-06; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Parkinson's Disease patients with genetic mutation
  Interventions: Diagnostic Test: Clinical examinations and clinical scales administration
- Control group: Parkinson's Disease patients without genetic mutation
  Interventions: Diagnostic Test: Clinical examinations and clinical scales administration

INTERVENTIONS:
Diagnostic Test: Clinical examinations and clinical scales administration — Psychometric assessment of cognitive and behavioral outcomes

SUMMARY:
The genetic landscape of Parkinson's disease (PD) is characterised by rare high penetrance pathogenic variants causing familial disease, genetic risk factor variants driving PD risk in a significant minority in PD cases and high frequency, low penetrance variants, which contribute a small increase of the risk of developing sporadic PD. This knowledge has the potential to have a major impact in the clinical care of people with PD.

The goal of this observational study is to evaluate the impact of genetic mutation on behavior and cognition in PD patients.

Patients will be assessed over time using test, questionnaire and standardised clinica scales. An initial assessment and annual follow-up assessments will be carried out for 5 years.

Researchers will compare data collected from patients with genetic mutation versus patients without mutation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Parkinson's Disease (PD)
* in use of dopaminergic medication (L-Dopa and/or dopamine agonists)
* genetic testing for mendelian forms of PD
* able to provide informed consent to participate in the study

Exclusion Criteria:

* Patients underwent Deep Brain Stimulation (DBS) treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants clinically diagnosed with Parkinson's Disease (PD) undergoing genetic testing for mendelian forms of PD
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2031-12-14 (Estimated); Study Completion 2031-12-14 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Annual assessments up to 5 years
  Cognitive impairment change from baseline until 5 years in Montreal Cognitive Assessment (MoCA; min. 0, max. 30, higher score means better outcome)
Beck Depression Inventory | Annual assessments up to 5 years
  Depressive symptoms change from baseline to 5 year (BDI-II, min 0, max 63, higher score means worse outcome)
State-Trait Anxiety Inventory | Annual assessments up to 5 years
  Anxiety symptoms change from baseline to 5 year (STAI, min 20, max 80, higher score means worse outcome)
Questionnaire for Impulsive-Compulsive Disorders in Parkinson | Annual assessments up to 5 years
  Impulsivity change from baseline to 5 years (QUIP, min 0, max 112, higher score means worse outcome)
Pittsburgh Sleep Quality Index | Annual assessments up to 5 years
  Sleep Quality change (PSQI, min 0, max 21, higher score means poorer sleep quality)
Parkinson's Disease Questionnaire-8 | Annual assessments up to 5 years
  Quality of life change from baseline to 5 years (PDQ-8, min 0, max 100, higher score means worse outcome)
Minnesota Multiphasic Personality Inventory 2-RF | Annual assessments up to 5 years
  Personality change from baseline to 5 years (MMPI-2-RF, cut-off: T>65 for clinical scales)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Mameli, Dr, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy